CLINICAL TRIAL: NCT03668652
Title: A Randomized Control Trial of Focal Prostate Ablation Versus Radical Prostatectomy
Brief Title: Focal Prostate Ablation Versus Radical Prostatectomy
Acronym: FARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Eduard Baco, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/703
Record Dates: First submitted 2018-04-15; First posted 2018-09-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; HIFU and TULSA Focal Treatment; Radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Masking Description: Focal treatment of prostate cancer using HIFU compared to Radical prostatectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal prostate cancer treatment by HIFU (Experimental): Patients with target lesion distance < 30 mm from the rectum will be treated with High Intensity Focused Ultrasound (HIFU) applied by FocalOne HIFU device and patients with lesion localized > 30 mm from the rectum will be treated with TULSA applied by TULSA-PRO device.
  Interventions: Device: Focal HIFU treatment using Focal One (EDAP TMS) or TULSA-PRO (Profound Medical)
- Radical Prostatectomy (Active Comparator): Robot assisted laparoscopic radical prostatectomy or open retro-pubic radical prostatectomy will be performed using validated radical prostatectomy technique. Nerve sparing surgery on side of cancer free prostate lobe will be performed and type of nerve sparing procedure will be specified.
  Interventions: Procedure: Radical prostatectomy

INTERVENTIONS:
Device: Focal HIFU treatment using Focal One (EDAP TMS) or TULSA-PRO (Profound Medical) — HIFU arm:
  Focal ablation of prostate cancer using HIFU Focal One or TULSA -PRO
  Arms: Focal prostate cancer treatment by HIFU
Procedure: Radical prostatectomy — Prostatectomy arm:
  Robot assisted or open retropubic prostatectomy
  Arms: Radical Prostatectomy

SUMMARY:
This study aims to compare the treatment results of HIFU and Radical prostatectomy.

DETAILED DESCRIPTION:
The FARP randomized control study will compare focal ablation of prostate using High Intensity Focused Ultrasound (HIFU) applied by FocalOne® or TULSA® device versus Radical Prostatectomy (RP) in patients with unilateral, intermediate risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Positive MRI (PIRAD 3-5) and biopsy proven unilateral prostate cancer classified as ISUP 1 (with cancer core length > 5mm) or ISUP 2-3 (any length) not eligible to active surveillance or watchful waiting
* PSA ≤ 20 ng/ml
* Treatment naive patients with localized prostate cancer (stage ≤ T2b)

Exclusion Criteria:

* Clinical stage T> 2b
* Metastatic lymph node on imaging
* Patients already treated for Pca (hormone therapy, EBRT)
* Patients with contra-indications to MRI
* Patients with active inflammatory bowel disease or previous rectal fistula
* History of previous pelvic radiotherapy
* History of bladder cancer
* History of bladder neck or urethral stricture
* Urogenital infection in progress
* Allergy to latex or gadolinium
* Patients on life support or suffering form unstable neurological diseases

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 213 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment failure. | At 36 months from the treatment date.
  Treatment failure in focal ablation arm is classified as the need for secondary whole gland treatment such as radical prostatectomy or EBRT due to detection of ISUP > 3 in treated and/or untreated areas on follow up prostate biopsy, or development of metastases on imaging.
  Treatment failure in the radical prostatectomy arm is classified as PSA > 0.2 ng/ml after surgery.

SECONDARY OUTCOMES:
Focal ablation failure. | Within 36 months from the treatment date.
  Focal ablation failure is classified as presence of Pca ISUP 1 ( > 5 mm) and/or ISUP 2-3 (any length) on follow up biopsies of the treated prostate zone.
Total re-ablation rate | Within 36 months from the treatment date.
  Secondary HIFU ablation was allowed if control biopsies revealed prostate cancer ISUP 1 ( > 5 mm) and/or ISUP 2-3) in treated or untreated areas.
Diagnostic failure. | Within 36 months from the treatment date.
  Diagnostic failure is classified as clinically significant cancer on control biopsy in the untreated area.
Cancer specific and all-cause mortality. | Within 36 months from the treatment date.
  Cause of the mortality will be evaluated and registered.
Difference in metastasis-free and overall survival. | Within 36 months years from the treatment date.
  Whole body MRI or PET CT will be performed if suspicion on metastases.
Difference in urinary continence between focal ablation and radical prostatectomy. | Within 36 months from the treatment date.
  Expanded Prostate Cancer Index Composite-26 (EPIC-26) questionnaire for the evaluation of continence will be used.
  Difference in pad free urinary continence and difference in number of pads needed per day.
  Difference in urinary incontinens defined as (full continence= 0 pads/day; security pad or mild incontinence = 1pad/day; moderate incontinence = 2pads/day and severe incontinence > 2pads/day).
Difference in erectile function between focal ablation and radical prostatectomy. | Within 36 months from the treatment date.
  International Index of Erectile Function (IIEF-5) questionnaire for the evaluation erectile function will be used.
  A score of 1-5 is awarded to each of the 5 questions. Change in total score will be measured between the baseline and most recent follow-up visit.
Difference in quality of life between focal ablation and radical prostatectomy. | Within 36 months from the treatment date.
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-c30) for the evaluation of quality of life between focal ablation and radical prostatectomy will be used.
Difference in adverse events related to both treatments. | Within 36 months from the treatment date
  All adverse events will be registered prospectively according to Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Baco, MD, PhD, Prof. assoc., Principal Investigator — Department of Cancer Surgery, Oslo University Hospital, Radiumhospitalet
Locations (1):
- Department of Cancer surgery, Oslo University Hospital, Radiumhospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
All data generated during this study will be evaluated at Oslo University Hospital